CLINICAL TRIAL: NCT02342262
Title: The Effects of Probiotics on the Frequency and Intensity of Migraine Attacks and Intestinal Permeability. A Placebo-controlled Trial
Brief Title: The Effect of Probiotics on the Frequency and Intensity of Migraine Attacks and Intestinal Permeability
Acronym: Promi2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL46401.081.13
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): EcologicBarrier, 5x10E9 cfu/day
  Interventions: Dietary Supplement: EcologicBarrier
- Placebo (Placebo Comparator): carrier material of Ecologic Barrier, not containing bacterial strains
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: EcologicBarrier — multispecies probiotic product, 2x10-9 cfu/gram
  Arms: Probiotics
Other: Placebo — similar appearance as the probiotic product, but without bacteria
  Arms: Placebo

SUMMARY:
RATIONALE: The prevalence of migraine is higher in patients with various intestinal diseases. An explanation could be that migraine is caused by a 'leaky gut': an increased intestinal permeability that allows food particles to pass the gastrointestinal wall. Probiotics may be able to improve intestinal barrier function.

OBJECTIVE: To test whether probiotics, as adjuvant therapy, can reduce incidence and severity of migraine attacks by reducing intestinal permeability.

STUDY DESIGN: 12-week placebo-controlled randomized double-blind intervention with selected probiotics.

STUDY POPULATION: Adults who experience at least 4 migraine attacks per month. INTERVENTION: Subjects will receive either one daily dose of 2 g of Ecologic® Barrier or 2 grams of the placebo, containing only the carrier material (both provided by Winclove Probiotics).

MAIN STUDY PARAMETERS/ENDPOINTS: Incidence and severity of migraine attacks, measured by diaries and validated headache questionnaires will be measured at baseline and after 4, 8, and 12 weeks of probiotic/placebo administration. Secondary, intestinal permeability will be measured by the lactulose/mannitol absorption test in urine (screening, baseline and 12 weeks) and by fecal zonulin (baseline, 4, 8, and 12 weeks). Inflammation will be assessed from blood C-reactive protein and cytokine concentrations (baseline, 4, 8, and 12 weeks). Fecal samples will also be used for microbial analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects confirm to have migraine characterized by :

  * Recurrent attacks of moderate to severe headaches, often one-sided and pounding, often with nausea and/or vomiting, aggravated by physical activity
  * Sensitivity for light or sounds is possible but not exclusive.
  * Attacks last for 4 to 72 hours.
* Self-reported frequency of migraine attacks (or days) at least 4 per month
* Fairly predictable/stable pattern of migraine attacks (frequency, duration, intensity)
* Age ≥ 18 years
* Good overall health (self-reported in medical questionnaire)

Exclusion Criteria:

* Migraine patients who suffer from chronic daily migraine/headaches
* Migraine patients who suffer from medication-dependent headaches
* Subjects who suffer from cluster headache or tension-type headaches
* Subjects who used antibiotics up to two months before the start of the study
* Subjects who are unwilling to stop taking probiotics other than study products
* Patients with a chronic use of non steroid anti inflammatory drugs (because of increased gut permeability)
* Patients with inflammatory bowel diseases (because of increased gut permeability)
* Pregnancy or lactation (because of their possible effect on migraine incidence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of migraine attacks | 12 weeks

SECONDARY OUTCOMES:
Intestinal permeability | 12 weeks
  Lactulose/mannitol in urine, zonulin in serum
Inflammation markers. | 12 weeks
  pro-inflammatory cytokines in serum

CONTACTS AND LOCATIONS:
Overall Officials: Nicole De Roos, PhD, Principal Investigator — Wageningen UR